CLINICAL TRIAL: NCT02775591
Title: Effect of Short-term Motilitone Therapy on Health-related Quality of Life in Parkinson's Disease Patients With Gastrointestinal Symptoms: a Multicenter, Double-blind Randomized, Placebo-controlled Trial
Brief Title: Effect of Short-term Motilitone Therapy on Health-related Quality of Life in PD Patients With Gastrointestinal Symptoms
Acronym: PASS-GI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Korea University Guro Hospital (Other); Hanyang University (Other); Seoul Veterans Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jee-Young Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26-2016-11
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease; Dyspepsia
MeSH Terms: conditions — Parkinson Disease; Dyspepsia | interventions — DA-9701

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motilitone arm (Experimental): DA-9701 (Motilitone) 30mg 1T three times per day for 4+8 weeks
  Interventions: Drug: DA-9701
- Placebo arm (Placebo Comparator): DA-9701 placebo 30mg 1T three times per day for 4 weeks, DA-9701 (Motilitone) 30mg 1T three times per day for 8 weeks
  Interventions: Drug: DA-9701; Drug: DA-9701 placebo

INTERVENTIONS:
Drug: DA-9701 — DA-9701 30mg Tablet
  Other Names: Motilitone
Drug: DA-9701 placebo — Placebo pill manufactured to mask DA-9701 30mg Tablet
  Other Names: Motilitone placebo
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to determine whether DA-9701(Motilitone) is effective and safe for the treatment on health-related quality of life in Parkinson's disease (PD) patients with gastrointestinal symptoms.

DETAILED DESCRIPTION:
Gastrointestinal (GI) symptoms are frequently complained by PD patients. To improve their symptoms, prokinetics are often used in clinics. However, some prokinetics are dopamine receptor antagonist which can aggravate motor symptoms of PD patients or develop tardive dyskinesia when it affects dopamine receptors of the brain.

DA-9701 (Motilitone) is recently developed herbal medication which has both 5-HT4 agonism and D2 antagonism. Furthermore, it does not cross the blood brain barrier that can be safely used in PD patients. Hypothetically it has a potential to be a good choice for the treatment of GI symptoms of PD patients. However, there has been no study that evaluates its efficacy and safety by randomized clinical trials in PD patients.

This study will evaluate the efficacy and safety of DA-9701 in the double-blind placebo-controlled phase 1 (4 weeks), and the long-term safety of DA-9701 in the open-label phase 2 (8 weeks after phase 1).

ELIGIBILITY:
Inclusion Criteria:

* Subjects were enrolled voluntarily and understood the contents of this clinical trial.
* Male or female Parkinson disease (PD) patients between 50 and 80 years
* Subjects who had not received prokinetics (itopride, mosapride, Corydalis tuber, levosulpiride, domperidone, etc.) at least 2 months prior to baseline visit
* Subjects complained at least one symptom of the following that suggests abnormal bowel functions: anorexia, nausea, abdominal distension, dyspepsia, early satiety, dysphagia, foreign body sensation associated with a meal, symptoms of gastroesophageal reflux, constipation, and defecation problem.

Exclusion Criteria:

* History of a gastrointestinal operation
* Subjects with active gastrointestinal diseases under treatment of gastroenterology within 1 month
* Existence of clinically significant cognitive decline or K-Minimental Status Exam score 20 or less
* Subjects had depression or other psychiatric disorders treated with medications such as antidepressants or antipsychotics; mood tranquilizers, benzodiazepines, and sleep pills were permitted with fixed dose during a period of the clinical trial
* Subjects with severe active comorbidities which could interfere the quality of life of the patient
* Subjects with medical conditions which make difficult to be enrolled to the trial judged by clinicians
* Subjects with hypersensitivity or adverse event related to DA-9701 (Motilitone)
* Prior participation to other clinical trials within 3 months

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in the Nepean dyspepsia index-Korean version scores | 4 weeks
  The Nepean dyspepsia index is a tool to measure gastrointestinal symptoms

SECONDARY OUTCOMES:
Change in bowel movements per day assessed by a bowel habit questionnaire. | 4 weeks, 12 weeks
  Mean bowel movements per day of recent 1 week will be asked using the bowel habit questionnaire.
Change in frequency of early satiety per day assessed by a bowel habit questionnaire. | 4 weeks, 12 weeks
  Mean frequency of early satiety per day of recent 1 week will be asked using the bowel habit questionnaire. The frequency will be categorized as following: 0, no event; 1, once a day; 2, twice a day; 3, every meal.
Change in frequency of gastric fullness after a meal per day assessed by a bowel habit questionnaire. | 4 weeks, 12 weeks
  Mean frequency of gastric fullness after a meal per day of recent 1 week will be asked using the bowel habit questionnaire. The frequency will be categorized as following: 0, no event; 1, once a day; 2, twice a day; 3, every meal.
Change in severity of epigastric pain assessed by a bowel habit questionnaire. | 4 weeks, 12 weeks
  Existence and severity of epigastric pain of recent 1 week will be asked using the bowel habit questionnaire. The severity will be categorized as following: 0, no event; 1, mild; 2, moderate; 3, severe; 4, very severe.
Change in the Bristol stool scale score | 4 weeks, 12 weeks
  This is a descriptive picture plate which patients can choose the type of their stool
Change in the Unified Parkinson's disease rating scale (UPDRS) scores | 4 weeks, 12 weeks
  This is a measure of the severity of Parkinson's disease
Change in the Parkinson's disease quality of life scale (PDQ-39) scores | 4 weeks, 12 weeks
  This is a measure of everyday quality of life affected by Parkinson's disease
Change in the Patient global improvement (PGI) scores | 4 weeks, 12 weeks
  This is a measure of patients perception of change in their gastrointestinal symptoms
Change in the Clinician global improvement (CGI) scores | 4 weeks, 12 weeks
  This is a measure of clinican's assessment of global clinical status of the patient
Change in the Nepean dyspepsia index-Korean version scores | 12 weeks
  This is a measure of changes in gastrointestinal symptoms at the end of this trial

CONTACTS AND LOCATIONS:
Overall Officials: Jee-Young Lee, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (5):
- South Korea (5):
  - Hanyang University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Veterans Healthcare Service Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
DATA including IPD can be shared individually upon request by qualified investigators excluding patients' personal information
Time Frame: The information will be judged by the principal investigator upon individual request.
Access Criteria: The information will be judged by the principal investigator upon individual request.

REFERENCES:
- [Derived] Choi JH, Lee JY, Cho JW, Koh SB, Yang YS, Yoo D, Shin CM, Kim HT. Double-Blind, Randomized, Placebo-Controlled Trial of DA-9701 in Parkinson's Disease: PASS-GI Study. Mov Disord. 2020 Nov;35(11):1966-1976. doi: 10.1002/mds.28219. Epub 2020 Aug 6. PMID 32761955